CLINICAL TRIAL: NCT01964469
Title: Consumer Access to Personal Health Information for Asthma Self-Management Phase 2 (Pilot Implementation)
Brief Title: Consumer Access to Personal Health Information for Asthma Self-Management
Acronym: ASMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Lung Association (Other); Ontario Ministry of Health and Long Term Care (Other Government); TELUS (Unknown); Canada Health Infoway (Other)
Responsible Party: Principal Investigator, Chris Licskai, Associate Professor of Medicine, University of Western Ontario, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00000940
Record Dates: First submitted 2013-01-21; First posted 2013-10-17 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Written self-management action plan (Placebo Comparator): Usual Care: Evidence-based best practice within the primary care asthma program including written self-management action plan and regular clinical review.
  Interventions: Behavioral: mobile & web-based action plan
- mobile & web based action plan (Experimental): Evidence-based best practice within the primary care asthma program, replacing the written action plan with the Breathe mobile health and web-based application.
  Interventions: Behavioral: mobile & web-based action plan
- Administrative data set (No Intervention): Health services use will be evaluated comparatively against our intervention population and our control and we will include health services utilization data from one year prior randomization.

INTERVENTIONS:
Behavioral: mobile & web-based action plan — Evidence-based best practice primary care asthma program including asthma self-management education replacing the written self-management action plan with the Breathe mobile health and web-based application
  Arms: Written self-management action plan; mobile & web based action plan

SUMMARY:
This study is to compare Smart phone mobile device and/or web based application asthma action plan to the standard of care paper based asthma action plan within an asthma program. The Primary hypothesis: Health Outcome - The Breathe mobile health and web-based application improves asthma related quality of life more than conventional best practice

DETAILED DESCRIPTION:
This study is a multi-centre, randomized controlled trial comparing a web-based (Smart phone mobile device, tablet and/or personal computer PC) asthma action plan application to best practice/usual care within an asthma program. A third external comparator arm will compare participants to all patients with asthma in Ontario using data obtained from the Ontario Asthma Surveillance Information System (OASIS) cohort, created from administrative data sets within the Institute for Clinical Evaluative Sciences (ICES). Subjects will be randomly assigned in blocks of four, stratified by site to, in a ratio of 1:1 intervention or control arms. The study will enrol approximately 400 patients in total at all study sites.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Age 18 of age or older
* Familiar with web technology
* Provide consent
* Understand/read/write English

Exclusion Criteria:

- Indication of other chronic lung diseases in the opinion of the physician that would impact their ability to participate in the trial or affect quality of life (Cystic Fibrosis, Chronic Obstructive Pulmonary Disease, Bronchiectasis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2013-02; Primary Completion 2014-06 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Health Outcome - Quality of Life | 6 months
  Health Outcome - The Breathe mobile health and web-based application improves asthma related quality of life more than conventional best practice.

SECONDARY OUTCOMES:
Quality - Health Care Utilization | 1 year
  Appropriateness of Care - Individuals with asthma who use the intervention will experience a decrease in the number of unplanned health system encounters

OTHER OUTCOMES:
Health Outcome - Quality | 1 year
  Improvements in symptom profile greater than conventional best practice.
Health Outcome - Quality of Life | 6 months
  Per protocol evaluation of the primary outcome, quality of life. It is anticipated that some subjects randomized to the intervention arm will not use the smartphone application. We seek to evaluate the primary outcome in those subjects who were adherent to the application compared to control subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Licskai, Principal Investigator — Lawson Health Research Institution
Locations (8):
- Canada (8):
  - Amherstburg FHT, Amherstburg, Ontario
  - Chatham-Kent FHT, Chatham, Ontario
  - Harrow FHT, Harrow, Ontario
  - Kingston Hospital Asthma Clinic, Kingston, Ontario
  - Leamington FHT, Leamington, Ontario
  - St. Joseph's Hospital Asthma Clinic, London, Ontario
  - Sault St. Marie Group Health Centre, Sault Ste. Marie, Ontario
  - Windsor FHT, Windsor, Ontario

REFERENCES:
- [Derived] Morita PP, Yeung MS, Ferrone M, Taite AK, Madeley C, Stevens Lavigne A, To T, Lougheed MD, Gupta S, Day AG, Cafazzo JA, Licskai C. A Patient-Centered Mobile Health System That Supports Asthma Self-Management (breathe): Design, Development, and Utilization. JMIR Mhealth Uhealth. 2019 Jan 28;7(1):e10956. doi: 10.2196/10956. PMID 30688654